CLINICAL TRIAL: NCT05778565
Title: Stretching of an Extraocular Rectus Muscle as a Weakening Procedure
Brief Title: Extraocular Muscle Stretching as a Weakening Procedure
Acronym: EOMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad Autonoma de Madrid (Other)
Responsible Party: Principal Investigator, Jaime Tejedor, Principal Investigator, Universidad Autonoma de Madrid
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OFTEOM-0322
Record Dates: First submitted 2023-02-20; First posted 2023-03-21 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Strabismus, Comitant
MeSH Terms: conditions — Strabismus

STUDY DESIGN:
Intervention Model Description: Extraocular muscle procedure
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Extraocular muscle stretching arm (Experimental)
  Interventions: Procedure: Extraocular muscle stretching

INTERVENTIONS:
Procedure: Extraocular muscle stretching — Extraocular muscle stretching to test its efficacy as a weakening procedure

SUMMARY:
Interventional case series. Non-operated patients with an indication of medial rectus muscle weakening surgery (deviation up to 20 PD) who could cooperate with topical or sub-Tenon's anesthesia. Clinical workup includes routine complete ophthalmological evaluation. One double needle 6/0 Mersilene suture is used on each side of the muscle at 4 mm distance of the insertion and pulled / stretched to insert in the sclera 3-5 mm posterior to the muscle locking passes.

Seven patients with esotropia of 12-20 PD were included.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring weakening of medial rectus muscle(s) for 12-20 PD of esotropia who could cooperate with topical / sub-Tenon's anesthesia, and had no previous eye muscle surgery

Exclusion Criteria:

* Patients with previous strabismus surgery

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2023-06-23 (Estimated); Study Completion 2023-06-23 (Estimated)

PRIMARY OUTCOMES:
Distance deviation at 2 months after surgery | 2 months
  Distance deviation at 2 months after surgery (alternate prim and cover)

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Tejedor, MD, PhD, Principal Investigator — Universite Abdou Moumouni de Niamey, Niger
Locations (1):
- UAM, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
When published

REFERENCES:
- [Derived] Tejedor J, Gutierrez-Carmona FJ. Extraocular Rectus Muscle Stretching as a Weakening Procedure. Ophthalmol Ther. 2023 Oct;12(5):2793-2800. doi: 10.1007/s40123-023-00756-3. Epub 2023 Jul 1. PMID 37392274